CLINICAL TRIAL: NCT03778151
Title: Repetitive TMS of the Precuneus: a Randomized Double-blinded Placebo-controlled Trial in Alzheimer's Disease Patients.
Brief Title: Repetitive TMS of the Default Mode Network in AD
Acronym: TMS-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giacomo Koch, Head of Laboratory, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC-2018
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRANSCRANIAL MAGNETIC STIMULATION (Active Comparator): repetitive TRANSCRANIAL MAGNETIC STIMULATION (rTMS) will be applied over the precuneus to modulate DMN activity. The rTMS treatment will consist of two phases: an intensive phase and a maintenance phase. The intensive phase will involve 2 weeks of treatment, 5 days per week (10 sessions, 1.600 pulses per day for a total of 16.000 pulses). The maintenance phase will consist of 1 session of treatment every week for 5 months (21 sessions, 100.800 pulses in total).
  Interventions: Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION
- SHAM TRANSCRANIAL MAGNETIC STIMULATION (Sham Comparator): SHAM TMS will be applied over the precuneus. The SHAM protocol will consist of two phases: an intensive phase and a maintenance phase. The intensive phase will involve 2 weeks of treatment, 5 days per week (10 sessions, 1.600 pulses per day for a total of 16.000 pulses). The maintenance phase will consist of 1 session of treatment every week for 5 months (21 sessions, 100.800 pulses in total).
  Interventions: Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION

INTERVENTIONS:
Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION — daily treatment session of REPETITIVE TRANSCRANIAL MAGNETIC STIMULATIO will be applied over precuneus for 20 minutes of consecutive blocks of 20Hz pulses for two seconds followed by 28 seconds of no stimulation.
  Other Names: RTMS

SUMMARY:
Alzheimer's disease is a global health challenge. Efforts aim at developing an effective treatment able to meet the needs of patients and their families. Thus, the primary aim of this project is to investigate the efficacy of a non-invasive brain stimulation, namely repetitive transcranial magnetic stimulation (rTMS), on cognition in patients with mild Alzheimer's disease. rTMS is considered a safe, well tolerated and relatively cheap treatment. The appealing idea of the intervention is to improve memory by directly modulating the activity of precuneus, key area linked to memory impairment. Patients will be treated with rTMS in two phases: an intensive phase and a maintenance phase for a total of six months. This project aims to provide a valid treatment to slow the worsening of symptoms and improve quality of life for those with Alzheimer's and their caregivers.

DETAILED DESCRIPTION:
Background: Alzheimer's disease (AD) is a neurodegenerative disorder characterized by severe disruption of large-scale brain networks connectivity. AD pathophysiology has been mainly associated with a breakdown of the Default Mode Network (DMN) and with a structural disconnection of parietal nodes. It has been shown that the precuneus (PC), a central hub of the DMN, is involved in successful episodic memory retrieval, working as a key area of the network activated by recognition memory. Recent anatomical works have shown that medial parietal regions are interconnected with the medial temporal region, which is implicated in memory retrieval. In particular, the PC was identified as a region demonstrating strong functional interconnectivity with the hippocampal formation. This is of particular relevance because PC is altered in AD. At early clinical stages of AD, PC is selectively vulnerable to early amyloid deposition, and plays a critical role in the conversion towards dementia.

Hypothesis: a novel therapeutic intervention for AD is repetitive Transcranial Magnetic Stimulation (rTMS). rTMS is a non- invasive approach that can be used to induce long lasting modulation of specific brain functions, inducing neuroplastic changes not only in the cortical site of stimulation, but also in remote interconnected areas. In a recent double blind randomized cross-over clinical pilot study, we found that a two-week course of daily high-frequency rTMS (20 Hz) treatment targeting the DMN (Stimulation site: PC) was able to induce an improvement in episodic memory compared to placebo. Indeed, TMS-EEG measurements showed that rTMS treatment, applied over the DMN, was capable to modulate the cortical activity in both the targeted areas (PC) as well as in functional connected regions of the DMN (Koch et al., 2018).

Specific aims: to investigate clinical efficacy and safety of DMN rTMS applied during 6 months in mild AD patients. To provide novel evidence that non-invasive treatment of network dysfunction, through stimulation of the PC, will represent an effective strategy to enhance cognitive functions and lead to substantial slowing of cognitive and functional decline in patients with mild AD. The findings yielded by the present project will have a potential strong impact on clinical practice of AD patients. Since rTMS is well tolerated and relatively low-priced, a positive result could lead to a fast application of the present proposal to the clinical experience. If successful, the proposed project will provide support for a novel treatment for cognitive dysfunction in AD patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient and the responsible caregiver have signed the Informed Consent Form.
2. The patient has probable AD, diagnosed according to NINCDS-ADRDA criteria.
3. The patient is a man or woman, aged ≤ 85 years.
4. The patient has a CDR total score of 0.5 or 1 (mild) and MMSE score of 18-26 (inclusive) at Screening.
5. Has at least one identified adult caregiver
6. The patient has been treated with acetylcholinesterase inhibitor (AChEI), i.e., donepezil, galantamine, or rivastigmine, at the time of Screening

   * For at least 3 months
   * The current dosage regimen must have remained stable for ≥ 8 weeks
   * It must be planned that the dosage regimen will remain stable throughout participation in the study
7. The patient is able to comply with the study procedures in the view of the investigator.

Exclusion Criteria:

1. Significant neurodegenerative disorder of the central nervous system other than Alzheimer's disease
2. Significant intracranial focal or vascular pathology seen on brain MRI scan
3. History of seizure (with the exception of febrile seizures in childhood)
4. Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM IV-TR) criteria met for any of the following within specified period:

   * Major depressive disorder (current)
   * Schizophrenia (lifetime)
   * Other psychotic disorders, bipolar disorder, or substance (including alcohol) related disorders (within the past 5 years)
5. Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MR imaging.
6. Treatment currently or within 3 months before Baseline with any of the following medications:

   * Typical and atypical antipsychotics (i.e. Clozapine, Olanzapine)
   * Antiepileptics drugs (i.e. Carbamazepine, Primidone, Pregabalin, Gabapentin)
   * Memantine

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating scale (CDR) sum of boxes | change from baseline to Week 24
  global cognition

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) | change from baseline to Week 24
  global cognition
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | change from baseline to Week 24
  functional activities
Neuropsychiatric Inventory (NPI) | change from baseline to Week 24
  behavioural symptoms
Frontal Assessment Battery (FAB) | change from baseline to Week 24
  frontal lobe functions
Immediate and delayed total recall score from the Rey Auditory Verbal Learning test (RAVLT) | change from baseline to Week 24
  memory
Cortical activity (TMS-EEG) | change from baseline to Week 24
  neurophysiological marker

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Motta, Study Director — Santa Lucia Foundation
Locations (2):
- Italy (2):
  - Giacomo Koch, Rome
  - Santa Lucia Foundation, Rome

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Koch G, Bonni S, Pellicciari MC, Casula EP, Mancini M, Esposito R, Ponzo V, Picazio S, Di Lorenzo F, Serra L, Motta C, Maiella M, Marra C, Cercignani M, Martorana A, Caltagirone C, Bozzali M. Transcranial magnetic stimulation of the precuneus enhances memory and neural activity in prodromal Alzheimer's disease. Neuroimage. 2018 Apr 1;169:302-311. doi: 10.1016/j.neuroimage.2017.12.048. Epub 2017 Dec 19. PMID 29277405
- [Background] Di Lorenzo F, Ponzo V, Bonni S, Motta C, Negrao Serra PC, Bozzali M, Caltagirone C, Martorana A, Koch G. Long-term potentiation-like cortical plasticity is disrupted in Alzheimer's disease patients independently from age of onset. Ann Neurol. 2016 Aug;80(2):202-10. doi: 10.1002/ana.24695. Epub 2016 Jul 8. PMID 27255833